CLINICAL TRIAL: NCT01435993
Title: A Randomized, Single Blind, Placebo-controlled, Single Ascending Dose/Repeat Dose Cohort Study to Assess Safety, Tolerability, Pharmacokinetics and Immunogenicity of GSK1223249 in Patients With Relapsing Forms of Multiple Sclerosis.
Brief Title: Multiple Doses of Anti-NOGO A in Relapsing Forms of Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114840; 2010-022664-12 (EudraCT Number)
Record Dates: First submitted 2011-08-25; First posted 2011-09-19 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Secondary-Progressive with relapses
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ozanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): GSK1223249 slow (60 minutes) intravenous infusion
  Interventions: Drug: GSK1223249
- Placebo (Placebo Comparator): Saline slow (60 minutes) intravenous infusion
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: GSK1223249 — Intravenous infusion
  Arms: Active
Other: Saline placebo — placebo intravenous infusion
  Arms: Placebo

SUMMARY:
This study will investigate an experimental new drug, GSK1223249 in patients diagnosed with relapsing forms of multiple sclerosis. The study will specifically investigate safety (vital signs like heart rate, blood pressure, Magnetic Resonance Imaging (MRI), and other markers of health from blood samples), tolerability (any side effects that occur, if any), and pharmacokinetics (how the body processes the drug and how long the drug stays in the blood, and in cerebro-spinal fluid). The study will also investigate if patients' own immune system interacts with GSK1223249.

DETAILED DESCRIPTION:
This study will be a randomised, placebo-controlled, single-blind (Investigator and Subject), single and repeat ascending dose protocol, in multiple sclerosis patients. The study is designed to evaluate the safety, tolerability, pharmacokinetics, and any potential for immunogenicity of GSK1223249 (a monoclonal antibody raised against Nogo-A), given intravenously in Multiple Sclerosis patients. The study will also evaluate exploratory endpoints including para-clinical activity via magnetic resonance imaging, cerebrospinal fluid pharmacokinetics, and effect of repeat dose administration of GSK1223249 on disability. Furthermore MS symptoms, such as relapses and individual symptom severity will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a relapsing form of MS .
* Using one of the following ongoing MS treatment strategies, defined as

  1. Currently receiving Beta-interferon/Copaxone for treatment of MS and have been receiving the current course of therapy for 3 or more months prior to screening, OR
  2. Not currently receiving disease modifying therapies for treatment of MS, and has not received such therapies for at least 3 months prior to screening.
* Demonstrated clinical activity in 2 years prior to screening, whilst receiving current/previous treatment regimen or prior to any treatment regimen
* Expanded Disability Status Scale (EDSS) score ≤6.0 at either the screening or baseline visit.
* Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* Body weight equal to or greater than: 50 kilogrammes

Exclusion Criteria:

* Complications/History of other diseases that may impact on safety of patients enroling into the study.
* Liver function test outside normal range for patient population
* Treatment with methylprednisolone or any other systemic steroid, for a relapse or otherwise, within 30 days of screening
* Treatment in the past 6 months with any of the following agents: Fingolimod (Gilenya), methotrexate, mitoxantrone, azathioprine, or other small molecule immunosuppressants.
* History of anaphilaxis to protein based therapeutics or mono-clonal antibodies.
* Positive result for Hapatitis B, HIV, and/or drugs of abuse, or excessive alcohol consumption.
* Not able to undergo MRI scanning safely, or Gadolinium (contrast enhancing agents) during MRI.
* Other significant infections e.g. Tuberculosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09-08 (Actual); Primary Completion 2012-01-23 (Actual); Study Completion 2012-01-23 (Actual)

PRIMARY OUTCOMES:
Safety | every 2-4 weeks over 7 months
  • Changes in vital signs, ECG monitoring, blood chemistry, haematology, urinalysis, monitoring of AEs and MS relapses (number, incidence, severity)

SECONDARY OUTCOMES:
Cmax values and AUC(0-∞) | Pre-dose; 1hr; 6hr; 12hr; 48hr; Day7; Day13; Follow-up
  Profile of Pharamcokinetics
Immunogenicity of GSK1223249 in MS patients | Predose; Day 85; Day169; Day197
  • Presence of antibodies to GSK1223249 to be assessed in serum samples using validated ECL assays.
Pharmacokinetics of GSK1223249 in cerebro-spinal fluid (CSF) in MS patients | Day7; or Day 29; or Day 35; or Day 85
  Measurement of GSK1223249 in CSF

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Verona, Veneto, Italy
- GSK Investigational Site, Lørenskog, Norway